CLINICAL TRIAL: NCT02659696
Title: An Observational Study to Evaluate the Efficacy of Nalfurafine Hydrochloride in Patients With Primary Biliary Cholangitis
Brief Title: Nalfurafine Hydrochloride for Pruritus in Patients With Primary Biliary Cholangitis
Status: Completed | Type: Observational
Sponsor: Teikyo University (Other)
Responsible Party: Principal Investigator, Atsushi Tanaka, Professor, Teikyo University
Other Study IDs: 15-037
Record Dates: First submitted 2015-12-19; First posted 2016-01-20 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Nalfurafine hydrochloride is a selective kappa-opioid receptor agonist developed in Japan, and in May 2015 the use of nalfurafine hydrochloride was officially approved in Japan for pruritus in patients with chronic liver diseases including PBC. In the current study, the investigators aimed to assess pruritus and overall QOL before and after administration of nalfurafine hydrochloride in patients with PBC. Furthermore, the investigators took serum sample from the enrolled patients and examine the association of pruritus with possible biomarkers.

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC, formally known as primary biliary cirrhosis) is a chronic cholestatic liver disease. Taking advantage of ursodeoxycholic acid (UDCA), the outcome of patients with PBC has been improved, comparable to those in general population. However, pruritus, which is often a persisting and annoying symptom, may decrease the quality of life (QOL) of patients with PBC. Although anti-histamines are administered for this the efficacy is limited, and no drugs which was clearly proved to be effective for suppressing pruritus have been developed worldwide.

Nalfurafine hydrochloride is a selective kappa-opioid receptor agonist developed in Japan, and in January 2009 approved for pruritus in patients with renal failure and under hemodialysis. A phase 3 trial of nalfurafine hydrochloride for pruritus in patients with chronic liver diseases was completed, indicating the efficacy as well as safety was confirmed. Therefore, in May 2015 the use of nalfurafine hydrochloride was officially approved in Japan for pruritus in patients with chronic liver diseases including PBC. However, only 59 patients with PBC were included and therefore it is still unclear whether nalfurafine chloride is effective in all PBC patients or a part of them, whether the effect of this drug depends on coadministered drugs or other complications, or whether this drug may improve QOL overall in patients with PBC.

In the current study, the investigators aimed to assess pruritus and overall QOL before and after administration of nalfurafine hydrochloride in patients with PBC, to answer the clinical questions described above. Furthermore, the investigators took serum sample from the enrolled patients and examine the association of pruritus with possible biomarkers.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of PBC
* Complain of moderate or severe pruritus
* Decided by physician to be administered nalfurafine hydrochloride

Exclusion criteria

* Severe liver damage (Child-Pugh grade C)
* Allergic to nalfurafine hydrochloride
* With no or mild pruritus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PBC, who complained of moderate or severe pruritus, and decided by physician to be administered nalfurafine hydrochloride
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with improvement of pruritus measured by PBC-40 | 3 months after administration of nalfurafine
  PBC-40 is a self-report questionnaire for the pruritus as well as health-related QOL in patients with PBC

SECONDARY OUTCOMES:
Proportion of patients with improvement of overall health-related QOL measured by PBC-40 | 3 months after administration of nalfurafine
  overall HRQOL is measured by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Tanaka, MD, PhD, Principal Investigator — Teikyo University
Locations (1):
- Teikyo University School of Medicine, Tokyo, Please Select, Japan

IPD SHARING:
Plan to Share IPD: No